CLINICAL TRIAL: NCT06274008
Title: Prospective Randomized Trial (RCT) of Adductor Canal Block With Bupivacaine Liposome Injectable Suspension (Exparel) for Anterior Cruciate Ligament Reconstruction vs. Standard Adductor Canal Block (ACB) With Bupivacaine
Brief Title: Exparel vs. ACB With Bupivacaine for ACL Reconstruction
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Children's Hospital of Orange County (Other)
Responsible Party: Principal Investigator, John Schlechter, Principal Investigator, Children's Hospital of Orange County
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 230110
Record Dates: First submitted 2023-11-03; First posted 2024-02-23 (Actual); Last update posted 2024-02-23 (Actual); Status verified 2024-02

CONDITIONS: ACL Tear; Opioid Misuse; Pain; Anxiety
MeSH Terms: conditions — Anterior Cruciate Ligament Injuries; Opioid-Related Disorders; Pain; Anxiety Disorders

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Exparel (Experimental): Adductor Canal Block with Bupivacaine Liposome Injectable Suspension Admixture bupivacaine 0.5 % 10 cc with Bupivacaine Liposome Injectable Suspension 10cc total 20
  Interventions: Drug: Exparel
- Standard ACB with bupivacaine (No Intervention): Standard Adductor Canal Block (ACB) with Bupivacaine Standardized amount of 0.5% bupivacaine 20 cc

INTERVENTIONS:
Drug: Exparel — Admixture bupivacaine 0.5 % 10 cc with Bupivacaine Liposome Injectable Suspension 10cc total 20
  Arms: Exparel

SUMMARY:
Opioid misuse and addiction among children and adolescents is an increasingly concerning problem. Post-surgical opioid prescriptions for commonly performed surgeries such as anterior cruciate ligament reconstruction (ACLR) increase opioid exposure in young athletes. The purpose of the current study is to determine if extended-release Bupivacaine Liposome Injectable Suspension (Exparel) is effective in decreasing at home narcotic consumption compared to standard Bupivacaine Adductor Canal Block for Anterior Cruciate Ligament (ACL) reconstruction/reconstruction for the surgical treatment of adolescents with ACL tears and concomitant pathology i.e. meniscus / cartilage injury/tear.

DETAILED DESCRIPTION:
Approximately 13% of high school seniors have reported nonmedical use of prescription opioids in their lifetimes with 8.7% to 11% reporting use within the last year. The second most common source of opioids (36.9%) in this population is leftover medication from previous legitimate prescriptions after injury or procedures. Before injury or surgery, most children and adolescents are narcotic naive. Medical use of opioids in this population increases the risk for nonmedical opioid misuse after high school by 33% (1). As orthopaedic surgeons, the surgeons are in a powerful position to understand and affect change in the adolescent population through patient/parent education and through controlling the amount and type of pain medications prescribed. The investigators propose a Double Blinded RCT of adolescents with ACL +/- meniscus tear to either bupivacaine ACB or Bupivacaine Liposome Injectable Suspension ACB (Exparel) to test whether injectable suspension reduces at home narcotic consumption postoperatively. Currently there is limited data available for the pediatric population and no known randomized controlled trials. Bupivacaine Liposome Injectable Suspension is FDA approved for use in adults but has been used in this pediatric population off-label for many years. Exparel is now FDA approved and indicated for single-dose infiltration in patients aged 6 years and older to produce postsurgical local analgesia. While widely used in the settings of a regional block in adolescents undergoing ACL reconstruction and other surgeries, it does not have specific FDA approval for the use in blocks. This is not uncommon practice and in fact many of the drugs used in pediatrics do not have specific approval by the FDA(2).

After enrollment, the research subject will be randomized into one of two arms and the anesthesiologist will be notified of the arm. Data will be collected at baseline, on day of surgery, and on days 1 through 14 postoperatively. Participants will be instructed to wear Actigraphs in the days leading up to surgery to obtain baseline sleep activity data.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are 7-17 years old undergoing elective ACL reconstruction/repair with American Society of Anesthesiologists (ASA) Classification 1-2 at Children's Hospital of Orange County (CHOC).
* Provision of signed and dated informed consent form
* Stated willingness to comply with all study procedures and availability for the duration of the study
* Surgery scheduled between the hours of 8am - 4pm

Exclusion Criteria:

* No prior major surgery (e.g. transplant procedures, cardiac, cranial surgeries)
* Learning disability or developmental delay. Learning disability or developmental delay will have been assessed by an outside specialist. Diagnosis will have either been communicated to attending physician by the patient or will be located in patient's medical record. Anything that would impede survey completion.

Ages: 7 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 96 (Estimated)
Dates: Start 2023-10-12 (Actual); Primary Completion 2024-10-30 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
At-home narcotic consumption by the patients as measured by the medication form completed by parents post discharge | Postoperative days 1-3, 7, and 14.
  Amount administered

SECONDARY OUTCOMES:
Postoperative pain level of child | Postoperative days 1-3, 7, and 14.
  Reported by parent and child via Visual Analogue Scale (VAS). Scores range from 0-100 with higher scores indicating more pain.
Functional disability of child | Baseline, Postoperative days 1-3, 7, and 14.
  The functional disability inventory is a measure of the degree to which children experience difficulty in physical and psychosocial functioning due to their physical health status. Respondents are asked to rate how much physical difficulty was perceived for a variety of everyday activities. Total scores are computed by summing the ratings for each item. Scores range from 0-60 with higher scores indicating greater perceived functional disability.
Parent and child anxiety | Baseline, Postoperative days 1-3, 7, and 14.
  The state questionnaire contains a 20-item, 4-point self-report rating scale for measuring anxiety. Total scores for situational anxiety range from 20 to 80; higher scores indicate higher levels of anxiety.
Child pain | Postoperative days 1-3, 7, and 14.
  The Parent's Postoperative Pain Measure is a 15-item measure to assess child's postoperative pain. Each item refers to an easily identifiable and specific behavior. Items are summed to yield a total score out of 15. A cutoff score of 6 identifies children who have clinically significant pain with excellent sensitivity and specificity.

CONTACTS AND LOCATIONS:
Locations (1):
- CHOC Children's Hospital, Orange, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] McCabe SE, West BT, Boyd CJ. Leftover prescription opioids and nonmedical use among high school seniors: a multi-cohort national study. J Adolesc Health. 2013 Apr;52(4):480-5. doi: 10.1016/j.jadohealth.2012.08.007. Epub 2012 Nov 22. PMID 23298996